CLINICAL TRIAL: NCT04687319
Title: Protocol for the Collection of Lung Mucus Samples From Care for a Rheology Research Programme
Brief Title: RHEology of the Pulmonary MUcus
Acronym: RHEMU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.298; 2020-A02367-32 (Other: ID RCB)
Record Dates: First submitted 2020-12-07; First posted 2020-12-29 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Bronchial Mucus in COPD and Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchial mucus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: bronchial mucus collection — mucus resulting from respiratory physiotherapy sessions for patients with cystic fibrosis or COPD, bronchial aspirations resulting from the bronchial fibroscopy programme

SUMMARY:
Patients for whom bronchial mucus collection has been performed as part of the treatment will be offered the opportunity to participate in the study.

* A rheology measurement will be carried out shortly after the collection of fresh bronchial mucus samples.
* Another part will be done on frozen bronchial mucus samples

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age.
* Patient consulting or hospitalised in the pneumology department and for whom an emission of bronchial mucus is planned as part of the treatment (mucus from respiratory physiotherapy sessions for patients with cystic fibrosis or COPD, bronchial aspirations from the bronchial fibroscopy programme).

Exclusion Criteria:

* Patient being opposed to the use of his mucus samples and data for this research.
* Patient protected by law (guardianship or curatorship), subject deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient consulting or hospitalised in the pneumology department and for whom an emission of bronchial mucus is planned as part of the treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of the rheology parameters studied | Day 1
  Establish operating protocols for obtaining reliable rheological measurements with a view to using them as biomarkers

IPD SHARING:
Plan to Share IPD: No